CLINICAL TRIAL: NCT05456373
Title: Intraoperative Use of ClearEdge Device in Breast Conserving Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LS BioPath (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSB-12345
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; lumpectomy; positive surgical margins
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision

STUDY DESIGN:
Intervention Model Description: multi-center, pivotal prospective, randomized clinical trial of the effect of imaging the excision specimen during surgical treatment of breast cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SoC+ClearEdge device - Standard of Care + study device (Experimental): Standard assessment of the surgical margins of the excised breast specimen during lumpectomy surgery plus the use of the study device to assess for breast cancer cells at the the margins
  Interventions: Device: ClearEdge device
- SoC - Standard of Care (No Intervention): Standard assessment of the surgical margins of the excised breast specimen during lumpectomy surgery

INTERVENTIONS:
Device: ClearEdge device — ClearEdge tissue imaging device uses a new technology to detect tissue abnormalities at the surgical margins of a surgically excised breast tissue specimen. Adding the use of the imaging device has the potential to assist the surgeon in identifying DCIS or invasive cancer involved margins of the excised specimen.
  Arms: SoC+ClearEdge device - Standard of Care + study device

SUMMARY:
Multi center, pivotal prospective, randomized clinical trial

The proposed randomized controlled study will evaluate the benefits of adding the ClearEdge imaging device to the Standard of Care (SoC) of margins assessment in breast conserving surgeries. The study will assess whether there is an improvement in the detection of DCIS or invasive cancer involved margins by measuring whether removal at the time of primary surgical treatment can reduce the need for repeat surgeries as compared to the SoC, which does not use the device.

DETAILED DESCRIPTION:
ClearEdge is a CE marked device already been used in several hospitals in the UK. It was used in a prospective single arm and 2 phases clinical study. It was demonstrated that surgeons successfully used the device to identify DCIS or invasive cancer involved margins and that it can reduce the need for repeat surgeries by meeting the margins depth criteria to require repeat operations. European Journal of Oncology Surgery. 2016; 42 (12): 1834-1840. In addition, the device was clinically evaluated by several hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are female (genotype)
2. Patients aged above 18 years, inclusive
3. Patients diagnosed with breast DCIS or invasive cancer recommended for lumpectomy procedure
4. Patients treated with neoadjuvant endocrine therapy may be enrolled

Exclusion Criteria:

1. Patients currently receiving chemotherapy
2. Patients having prior ipsilateral surgical treatment for breast cancer
3. Patients who have had radiation therapy for ipsilateral breast cancer or for other malignancy that includes breast tissue in the radiation field (e.g. Hodgkin's lymphoma)
4. Patients who have breast implants
5. Patients who are pregnant and/or lactating
6. Patients participating in other breast cancer studies involving surgical treatment to the breast in the past 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with positive margins post-op | In the operating room compared to pathology assessment within 1 week post-op
  The percentage of patients with DCIS or invasive cancer involved margins as determined by pathology PM after evaluation with SoC or SoC+ClearEdge.

SECONDARY OUTCOMES:
FN and FP rates | within weeks post-op
  The per-patient FN rate and FP rate for SoC compared to permanent section pathology

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Wong, MD, Principal Investigator — University of California, San Francisco Medical Center
Locations (1):
- UCSF Medical Center at Mission Bay, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Possibly to Study Site PIs